CLINICAL TRIAL: NCT01240291
Title: Effect of Intravenous GLutamine Supplementation IN Trauma Patients Receiving Enteral Nutrition Study Protocol (GLINT Study): A Prospective, Blinded, Randomized, Placebo-controlled Clinical Trial
Brief Title: The Clinical Role of Intravenous Glutamine in Trauma Patients Receiving Enteral Nutrition
Acronym: GLINT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Principal Investigator, Ruqaiya Al-Balushi, Researcher, Royal Brisbane and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC/10/QRBW/131
Record Dates: First submitted 2010-11-01; First posted 2010-11-15 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Trauma; Critically Ill
Keywords: glutamine; trauma; alanyl-glutamine
MeSH Terms: conditions — Multiple Trauma; Critical Illness; Wounds and Injuries | interventions — alanylglutamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- alanyl-glutamine (Experimental): Intravenous alanyl-glutamine (0.5 g/kg body weight/day)
  Interventions: Dietary Supplement: Dipeptiven
- normal saline (Placebo Comparator): Intravenous placebo (normal saline; 0.9 %)
  Interventions: Dietary Supplement: normal saline

INTERVENTIONS:
Dietary Supplement: Dipeptiven — Intravenous alanyl-glutamine (0.5 g/kg body weight; i.e. 0.35 g L-glutamine / kg body weight; continuous infusion (20-24 hr/day) via central venous access for a maximum duration of 3 weeks.
  Other Names: Fresenius Kabi
  Arms: alanyl-glutamine
Dietary Supplement: normal saline — 0.5 g/kg bod weight /day, continuous infusion (20-24 hr/day) via central venous access for a maximum duration of 3 weeks
  Other Names: NaCl
  Arms: normal saline

SUMMARY:
The purpose of this trial is to investigate if pharmacologically safe dose intravenous glutamine dipeptide supplementation to multiple trauma patients receiving enteral nutrition is associated with improved clinical outcomes in terms of decreased organ dysfunction, infectious complications, and other secondary outcomes

DETAILED DESCRIPTION:
Trauma Patients are characterized by alteration in the immune response, increased exposure to infectious complications, sepsis, and consequently organ failure and death. Glutamine supplementation to parenteral nutrition is one of the nutritional interventions that have been proven to be associated with improved survival rate, decreased infectious morbidity, costs, intensive care unit, and hospital length of stay. However, glutamine supplementation in patients receiving enteral nutrition and its best route are still controversial. A number of trials investigated the beneficial effects of intravenous alanyl-glutamine supplementation in critically ill patients receiving enteral nutrition. However, these trials were: pilot trials, investigated surrogate outcomes, or supplementation was for a short period of time. Therefore, a well designed trial is needed to investigate the effect of intravenous alanyl-glutamine supplementation in critically ill patients with multiple trauma receiving enteral nutrition on major clinical outcomes.

Our hypothesis is that trauma patients receiving standard enteral nutrition supplemented with intravenous alanyl-glutamine will demonstrate improved clinical outcomes compared to patients receiving standard enteral nutrition without supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-58 years
* Patients admitted with a diagnosis of multiple trauma requiring enteral feeding for > 48 hours
* Expected length of stay in ICU > 48 hours
* Has a functional access for enteral tube feeding and a central access for administration of test solution
* Negative Beta HCG (pregnancy test) in females (18-60 years)

Exclusion Criteria:

* Age < 18 years
* Significant hepatic failure (Patients with Childs C Cirrhosis)
* Severe renal failure (estimated glomerular filtration rate [eGFR] < 50 ml/min)
* Patients with severe metabolic acidosis (pH <7.35)
* Not expected to be in the ICU > 48 hours (due to imminent death)
* Unable to tolerate enteral nutrition within 72 hours
* Enrolment in other ICU intervention study if contraindicated
* Patients in whom parenteral nutrition is required from the outset
* Absolute contraindication to enteral nutrition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The change in daily total Sequential Organ Failure Assessment Score (SOFA)each day over 10 days. | daily until discharge from intensive care unit, death or maximum duration of 10 days.
  The change in daily total SOFA score plotted each day over 10 days, where we will compare the regression slope between the two arms of the study.

SECONDARY OUTCOMES:
The change in daily total Sequential Organ failure Assessment Score (SOFA) on the last day of treatment as a measure of severity of organ dysfunction. | Last day of treatment
Number of infections that are documented during intensive care unit stay. | During intensive care unit stay.
Number of deaths occuring on or before day 60. | within 60 days.
Length of stay in intensive care unit. | At discharge from intensive care unit.
Length of stay in hospital. | At hospital discharge.
  Length of stay in hospital (if delayed discharge due to placement problems, will record from the date the patient is regarded as fit for discharge by medical staff).
Number of days on mechanical ventilation. | during intensive care unit stay.
Number of days of antibiotic use during intensive care unit stay. | during intensive care unit stay.
Fat free mass and fat percentage as a measure of body composition by Bioelectric Impedance analysis (BIA). | every 2 days until discharge from the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lipman, MBBCh, MD, Principal Investigator — Royal Brisbane & Women's Hpsoital
Locations (1):
- Royal Brisbane & Women's Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Al Balushi RM, Paratz JD, Cohen J, Banks M, Dulhunty J, Roberts JA, Lipman J. Effect of intravenous GLutamine supplementation IN Trauma patients receiving enteral nutrition study protocol (GLINT Study): a prospective, blinded, randomised, placebo-controlled clinical trial. BMJ Open. 2011 Nov 14;1(2):e000334. doi: 10.1136/bmjopen-2011-000334. Print 2011. PMID 22102646